CLINICAL TRIAL: NCT02156596
Title: Intravenous Treatment With Non Steroidal Anti Inflammatory Drugs (NSAID) Versus Nebulized Morphine (NM) Analgesia for First-line Renal Colic: Randomized Controlled Double-blind Single-center Study.
Brief Title: IV NSAI Versus Nebulized Morphine Analgesia for First-line Renal Colic
Acronym: NSAIvsNM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Clinical Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSAI vs Morphine
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Renal Colic
Keywords: renal colic; nebulised morphine; Intravenous NSAID
MeSH Terms: conditions — Renal Colic | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous NSAI (Active Comparator): patients received 100 mg of ketoprofen (NSAID) by IV root and in parallel 3 nebulisation of serum saline (SS) over 30 minutes.
  Interventions: Drug: IV NSAI; Drug: Nebulised Serum Saline
- Nebulised Morphine (Experimental): patients received 3 nebulisation of morphine (5 mg each) and in parallel 50 ml of SS by IV root over 30 minutes.
  Interventions: Drug: NM; Drug: IV Serum Saline

INTERVENTIONS:
Drug: IV NSAI — 100 mg of ketoprofen in 50 ml volume given in 30 minutes by IV root
  Other Names: ketoprofen IV
  Arms: Intravenous NSAI
Drug: NM — 3 nebulisations of 5 mg morphine chlorhydrate each given over 30 minutes (10 minutes per nebulisation)
  Other Names: morphine
  Arms: Nebulised Morphine
Drug: IV Serum Saline — 50 ml of SS is given by IV root over 30 minutes
  Other Names: serum saline
  Arms: Nebulised Morphine
Drug: Nebulised Serum Saline — 3 nebulisations of 5ml SS each are given over 30 minutes
  Other Names: serum saline
  Arms: Intravenous NSAI

SUMMARY:
The aim of the investigators study was to evaluate the feasibility, efficacy and safety of nebulized morphine compared with non-steroidal anti-inflammatory (NSAI)intravenously in the management of renal colic.

Determine the need for systematic outpatient prescription of NSAI.

DETAILED DESCRIPTION:
Renal colic are a frequent cause of consultation in the emergency departement (ED).

They count for approximatively 20% of patients presenting to the ED with severe acute onset abdominal pain.

For acute treatment of renal colics (RC), guidelines recommend the use of intravenous (IV) non-steroidal anti-inflammatory (NSAI) drugs in association with antalgics like Paracetamol or Morphine.

But the NSAID present many inconvenient and cannot be used in some type of patients; that's why the investigators investigated the use of other drugs, such as nebulised morphine, in the ED treatment of renal colics.

the NM has the adequacy of being quickest, more practical to use and more tolerated than the IV NSAID.

In this study, the investigators aim to assess the feasibility, efficacity and safety of nebulised morphine compared to intravenous NSAID in the treatment of RC.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years old
* Consenting to participate in the study
* Diagnosis of renal colic matching flank pain / lumbar fossa sided with dipstick and / or imaging confirmed the diagnosis
* VAS> 50% at consultation

Exclusion Criteria:

* Inability to assess pain VAS;
* Pregnant or lactating woman;
* Recognized renal disease (glomerular filtration rate <60ml/kg/1.73m2);
* Known hepatic insufficiency;
* Known or suspected allergy to NSAIDs, morphine
* Peptic ulcer known;

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
efficacity: VAS pain reduction | 5, 15, 30, 45 and 60 minutes
  The effectiveness of treatment is defined by a decrease in the intensity of pain corresponding to a decrease of the VAS above 50% at 60 minutes compared to baseline.

SECONDARY OUTCOMES:
feasibility of the study: number of patients accepting the adhesion to protocol | at base line and at 60 minutes
  the feasibility is assessed by comparing the number of patients accepting the protocol to the total number of patients consulting for RC; and the number of patients that actually completed the protocol course (if above 50%, the protocol is considered feasable).
safety: side effects of treatment | 5, 15, 30, 45 and 60 minutes
  the safety of treatment is evaluated by the occurence of side effects at any time of the protocol.
  only major side effects (repeated vomiting, untolerated dizziness, conscience troubles, dyspnea and allergic reaction) are admitted to stop the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (1):
- Hospital of Fattouma Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official department site — http://www.urgencemonastir.com